CLINICAL TRIAL: NCT00361140
Title: Busulfan Dose Escalation Study Based on AUC in the Setting of Busulfan/Fludarabine Conditioning Prior to Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Busulfan Safety/Efficacy as Conditioning Prior to Hematopoietic Cell Transplantation (HCT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14178
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2013-06

CONDITIONS: Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Lymphocytic; Myeloma; Lymphoma
Keywords: Busulfan; Fludarabine; Chimerism; Allogeneic stem cell transplantation (HCT); Myelodysplastic Syndromes; Leukemia Myeloproliferative disorders (MPD); Leukemia, Lymphocytic; Myeloma; Lymphoma; AUC; Hematologic malignancies
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Lymphoid; Neoplasms, Plasma Cell; Lymphoma; Hematologic Neoplasms | interventions — Busulfan; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AUC 6000 (Experimental): Busulfan AUC Level 1: 6000 +/- 600 uM-min
  Fludarabine 40mg/m2 IV over 1 hour
  Interventions: Drug: Busulfan; Drug: Fludarabine
- AUC 7500 (Experimental): Busulfan AUC Level 2: 7500 +/- 750 uM-min
  Fludarabine 40mg/m2 IV over 1 hour
  Interventions: Drug: Busulfan; Drug: Fludarabine
- AUC 9000 (Experimental): AUC Level 3: 9000 +/- 900 uM-min
  Fludarabine 40mg/m2 IV over 1 hour
  Interventions: Drug: Busulfan; Drug: Fludarabine

INTERVENTIONS:
Drug: Busulfan — Bu IV (BusulfexR) over 3 hours on days -6, -5, -4, and -3. Day -6 and -5 doses for patients on Level 1 will be 170mg/m2. This dose is based on the dose used by DeLima (2004) adjusted proportionately to achieve an AUC of 6000uM-min. Subsequent daily doses for patients on Level 1 will be adjusted to achieve an average AUC of 6000uM-min.
  Day -6 and -5 doses for patients on Level 2 will be based on the mean dose required on Level 1 to achieve target AUC then adjusted proportionally for new target AUC.
  Subsequent daily doses will be adjusted to achieve target AUCs.
  Other Names: Busulfex(R)
Drug: Fludarabine — Fludarabine 40mg/m2 IV over 1 hour on days -6, -5, -4, and -3
  Other Names: Fludarabine Phosphate

SUMMARY:
Pre-transplant conditioning will include Fludarabine and dose-escalated Busulfan on days -6, -5, -4, and -3. Daily treatment doses will be adjusted to achieve target area under the plasma concentration time curve (AUC). Day 0 is the day of hematopoietic progenitor cell reinfusion. Supportive care will be based on institutional guidelines. Blood samples will be collected for dose modification based on the AUC levels. Dose escalation will proceed to determine the maximally tolerated level or AUC to evaluate the potential therapeutic benefit of higher doses of busulfan.

DETAILED DESCRIPTION:
Patients will receive anti-seizure prophylaxis beginning on day -7. Pre-transplant conditioning will include Fludarabine and dose-escalated Busulfan on days -6, -5, -4, and -3. Daily treatment doses will be adjusted to achieve target AUCs (area under the plasma concentration time curve). Day 0 is the day of hematopoietic progenitor cell reinfusion.

Supportive care will be based on institutional guidelines. In an effort to prevent hepatotoxicity, ursodiol will be given to patients. During chemotherapy patients will not receive concurrent metronidazole, itraconazole, or be given acetaminophen.

Blood samples will be collected at specific times after Dose 1 and Dose 4 and dose modification will be determined or based on the desired AUC levels. Doses 3 and/or 4 will be adjusted to achieve an average daily Busulfan AUC over the 4 treatment days.

Dose escalation will proceed through 3 dose levels to determine the maximally tolerated level or AUC to evaluate the potential therapeutic benefit of higher doses of busulfan.

Graft assessment, processing, and characterization will be done as per institutional guidelines. Donor-recipient chimerism (two genetically distinct types of blood cells) will be characterized by samples obtained pre-transplant and on days 30+/- 7, 90+/-7 and 360+/-30 post-transplant.

ELIGIBILITY:
Inclusion Criteria - Recipient:

* HLA A, B, C, DRB1 8/8 or 7/8 matched related or unrelated donor. HLA-DQ mismatches are not considered ie they are allowed in addition to these.
* Histologically confirmed diagnosis by pathologic review
* Diagnosis of any of the following:

  1. Acute myelogenous leukemia (AML), Acute lymphoblastic leukemia (ALL), or Non-Hodgkin's Leukemia (NHL), in first remission with high risk of relapse, refractory to primary chemotherapy, or after first relapse; acute biphenotypic or undifferentiated leukemia is also included
  2. Myelodysplastic Syndrome (MDS), with IPSS >1
  3. Chronic myelogenous leukemia (CML), with GleevecR-refractory or intolerant chronic phase, or beyond chronic phase by morphology or cytogenetics
  4. Myeloproliferative disorders, including Ph-negative CML, myelofibrosis and chronic myelomonocytic leukemia (CMML)
  5. Multiple myeloma, refractory to two or more lines of therapy.
  6. Chronic lymphocytic leukemia (CLL), refractory to fludarabine
  7. Hodgkin's disease, refractory to primary chemotherapy or after first relapse
  8. Karnofsky performance status 70-100%
* Organ function:

  1. Pulmonary: Diffusing capacity of lung for carbon monoxide (DLCO) greater than 50%
  2. Cardiac: Left ventricular ejection fraction greater than 45%
  3. Renal: Creatinine clearance (measured or calculated) equal or greater than 50 ml/min
  4. Hepatic: Total bilirubin less than or equal to 2 mg/dL, (Gilbert and other syndromes with increased indirect bilirubin should be allowed); serum transaminases less than two times the upper limit of normal.
* Signed informed consent form in accordance with institutional policies

Exclusion Criteria - Recipient:

* Pregnant or lactating women
* HIV or seropositive, confirmed by nucleic acid test (NAT)
* Active central nervous system (CNS) malignancy
* Patients with current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings) are ineligible.
* Unfavorable psychosocial evaluation or history of poor compliance to prescribed medical care
* Current use of metronidazole or acetominophen, unless medically necessary; patients must discontinue use of these agents at least 7 days prior to the start of BusulfexR administration
* Prior use of MylotargR (gemtuzumab ozogamicin)
* Prior Hematopoietic Cell Transplantation (HCT)
* Prior chest or abdominal irradiation with greater than 1800 cGy
* Presence of any of the following comorbid conditions:

  1. History of myocardial infarction or coronary artery disease requiring catheterization or stent placements less than six months prior to enrollment. All participants with history of myocardial infarction or coronary artery disease must have clearance by a cardiologist to be enrolled.
  2. Congestive heart failure (even if symptomatically controlled)
  3. Peripheral vascular disease (including intermittent claudication or history of bypass for arterial insufficiency)
  4. Untreated thoracic or abdominal aneurysm (6 cm or more)
  5. History of any cerebrovascular accident including transient ischemic attacks
  6. Dementia
  7. Connective tissue/rheumatologic disorders with active disease
  8. Diabetes uncontrolled by medication (including insulin)
  9. Hemiplegia/paraplegia
  10. History of prior malignancy (excluding nonmelanoma skin or cervical carcinoma after curative resection) less than 5 years from enrollment with the following exception. Cancer treated with curative intent less than 5 years will be reviewed on a case-by-case basis by the Principal Investigator.
  11. History of renal failure requiring renal replacement therapy (e.g., hemodialysis, peritoneal dialysis, etc.)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Field, PhD, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Janelle Perkins, PharmD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Result] Perkins JB, Kim J, Anasetti C, Fernandez HF, Perez LE, Ayala E, Kharfan-Dabaja MA, Tomblyn MR, Sullivan DM, Pidala JA, Field TL. Maximally tolerated busulfan systemic exposure in combination with fludarabine as conditioning before allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2012 Jul;18(7):1099-107. doi: 10.1016/j.bbmt.2011.12.584. Epub 2011 Dec 23. PMID 22198540
- See also: Moffitt Cancer Center Clinical Trials website — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: BMT population recruited from 08/01/2005 through 09/09/2012
Pre-assignment Details: candidates not meeting eligibility criteria excluded.
Groups:
- AUC Level 1: Busulfan targeted area under the curve, level 1: 6000 +/- 600 uM-min
- AUC Level 2: Busulfan targeted area under the curve, level 2: 7500 +/- 750 uM-min
- AUC Level 3: Busulfan targeted area under the curve, level 3: 9000 +/- 900 uM-min
Period: Overall Study
Arm/Group | AUC Level 1 | AUC Level 2 | AUC Level 3
Started | 40 | 29 | 3
Completed | 40 | 29 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AUC Level 1 | AUC Level 2 | AUC Level 3 | Total
Number analyzed (Participants) | 40 | 29 | 3 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 29 | 3 | 72
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 3 | 36
  Male | 24 | 12 | 0 | 36
Region of Enrollment [Number; unit: participants]
  United States | 40 | 29 | 3 | 72

OUTCOME MEASURES:

1. Secondary Outcome: Severe Venous Occlusive Disease (VOD)/ Sinusoidal Obstructive Syndrome (SOS)
Description: The number of subjects with severe VOD / SOS; severity staged according to criteria set forth by McDonald G.B., Hinds M.S., Fisher L.D., et al. Veno-occlusive disease of the liver and multiorgan failure after bone marrow transplantation: a cohort study of 355 patients. Ann Intern Med. 1993;118:255-267. Assessed within the first 100 days post transplant.
Time Frame: 100 days
Population: Intent to treat
Measure: Number; unit: participants
Groups:
- AUC 6000: Busulfan AUC Level 1: 6000 +/- 600 uM-min Fludarabine 40 mg/m^2 I.V. over 1 hour
- AUC 7500: Busulfan AUC Level 2: 7500 +/- 750 uM-min Fludarabine 40 mg/m^2 I.V. over 1 hour
- AUC 9000: Busulfan AUC Level 3: 9000 +/- 900 uM-min Fludarabine 40 mg/m^2 I.V. over 1 hour
Arm/Group | AUC 6000 | AUC 7500 | AUC 9000
Number analyzed (Participants) | 40 | 29 | 3
participants | 0 | 1 | 2
Statistical Analysis 1: Comparison: AUC 6000 vs AUC 7500 vs AUC 9000; Test type: Superiority or Other; p = .007, Chi-squared

2. Primary Outcome: Non-relapse Mortality
Description: The number of participants dead due to causes unrelated to relapse within the first 100 days post transplant.
Time Frame: 100 days
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | AUC 6000 | AUC 7500 | AUC 9000
Number analyzed (Participants) | 40 | 29 | 3
participants | 3 | 4 | 2
Statistical Analysis 1: Comparison: AUC 6000 vs AUC 7500 vs AUC 9000; Sample size: dependent on dose escalation. Once the maximum tolerated dose (MTD) is reached, a total of 30 patients will be accrued to that level. If maximally tolerated AUC is level 1, a total of 30 patients will be treated on this level using tacrolimus and methotrexate as GVHD prophylaxis. This will provide 95% confidence intervals for 100-day non-relapse mortality and non-fatal toxicities with ½ widths not exceeding 0.18. Hazard ratios were calculated per the method of Gray (reference given); Test type: Superiority or Other; p = .07, Gray; Gray RJ. A class of K-sample tests for comparing the cumulative incidence of a competing risk. Ann Stat. 1988;16:1141-1154; Hazard Ratio (HR) = 6.27, 95% CI 2-sided [0.92 to 42.48]

ADVERSE EVENTS:
Description: Anticipated "other than serious" Allogeneic Hematopoietic Cell Transplantation (HCT) adverse events were not tabulated.
Arm/Group | AUC Level 1 | AUC Level 2 | AUC Level 3
Serious Adverse Events (participants affected / at risk) | 2/40 | 13/29 | 2/3
Other Adverse Events (participants affected / at risk) | 0/40 | 0/29 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUC Level 1 (N=40) | AUC Level 2 (N=29) | AUC Level 3 (N=3)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Unlikely to be related
Hemorrhage, GI - Stomach (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — Unlikely to be related
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Unlikely to be related
Death not associated with CTCAE term - Death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Hepatobiliary/Pancreas - Other, VOD (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) — Unrelated
Infection with normal ANC or Grade 1 or 2 neutrophils - Stomach (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Unrelated
AST, SGOT - high (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Mental status (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Pulmonary/Upper Respiratory - Other, edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No